CLINICAL TRIAL: NCT02691455
Title: The AGS Second Aqueous Shunt Implant vs. Transscleral Cyclophotocoagulation Treatment Study
Brief Title: The American Glaucoma Society (AGS) Second Aqueous Shunt Implant vs. Transscleral Cyclophotocoagulation Treatment Study (ASSISTS)
Acronym: ASSISTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting participants
Sponsor: Robert Feldman (Other)
Responsible Party: Sponsor-Investigator, Robert Feldman, M.D., The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-15-1053
Record Dates: First submitted 2016-02-15; First posted 2016-02-25 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Second Aqueous Shunt (Active Comparator): Second Aqueous Shunt
  Either a Baerveldt Glaucoma Implant 350-mm2 BG101-350 or an Ahmed Model FP7 Flexible Plate must be used for all participants unless there is insufficient space, in which case a Baerveldt Glaucoma Implant 250-mm2 BG103-250 may be used.
  Interventions: Device: Baerveldt Glaucoma Implant 350-mm2 / BG101-350; Device: Ahmed Model FP7 Flexible Plate; Device: Baerveldt Glaucoma Implant 250-mm2 / BG103-250
- Transscleral Cyclophotocoagulation (Active Comparator): Transscleral Diode Laser Cyclophotocoagulation
  Interventions: Procedure: Transscleral Diode Laser Cyclophotocoagulation

INTERVENTIONS:
Device: Baerveldt Glaucoma Implant 350-mm2 / BG101-350
  Arms: Second Aqueous Shunt
Procedure: Transscleral Diode Laser Cyclophotocoagulation — Recommended setting are 2000 milliwatt (mW) for 2 seconds, 1850 mW for 3 seconds or 1750 mW for 4 second duration, titrating the energy up or down just below where a pop is heard.
  Other Names: Transscleral Diode Laser Cyclophotocoagulation (TLC)
  Arms: Transscleral Cyclophotocoagulation
Device: Ahmed Model FP7 Flexible Plate
  Arms: Second Aqueous Shunt
Device: Baerveldt Glaucoma Implant 250-mm2 / BG103-250
  Arms: Second Aqueous Shunt

SUMMARY:
Outcomes of subjects with uncontrolled glaucoma with a single existing aqueous tube shunt implant undergoing a second aqueous shunt to transscleral diode laser cyclophotocoagulation.

DETAILED DESCRIPTION:
This is a study comparing short- (1 year), mid- (3 years), and long-term (5 years) cumulative incidences of failures in participants who undergo a second aqueous shunt (SAS) to those cumulative incidences of failures in participants who undergo a second aqueous shunt (SAS) to those cumulative incidences of failures in participants who undergo transscleral diode laser cyclophotocoagulation (TLC) for eyes with uncontrolled glaucoma with a single existing aqueous tube shunt procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18 to 85 years of age
* Glaucoma not adequately controlled (IOP >18 mmHg on maximum tolerated topical therapy) with a single aqueous shunt (AS).
* Best-corrected visual acuity (BCVA) of hand motion (HM) or better in the study eye

Exclusion Criteria:

* Monocular
* Presence of more than one AS in the study eye
* Previous cyclodestruction in the study eye
* Presence of active iris neovascularization in the study eye
* Binocular diplopia
* Presence of scleral buckle in the study eye
* History or scleritis in either eye
* History of scleromalacia in the study eye
* Insufficient conjunctiva to cover AS in the study eye
* IOP cannot be accurately measured with Goldmann applanation, Pneumotonometry, or Tono-Pen in the study eye
* Presence of silicone oil in the study eye
* Presence of retinal detachment in the study eye
* Presence of intraocular or orbital tumor affecting the study eye
* Need for cataract extraction or concurrent procedure at the time of study treatment, except tectonic aqueous shunt revisions for both groups is allowed.
* In the opinion of the investigator, should not be enrolled in this study
* Unwilling or unable to give consent and satisfy requirements of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldman, MD, Study Chair — Robert Cizik Eye Clinic
Locations (23):
- United States (23):
  - University of California San Diego - Shiley Eye Institute, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Bascom Palmer Eye Institute - Miami, Miami, Florida
  - Bascom Palmer Eye Institute, Palm Beach Gardens, Florida
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Stiles Eyecare Excellence and Glaucoma Institute, Overland Park, Kansas
  - New England Eye Center - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Glaucoma Consultants of St. Louis, Chesterfield, Missouri
  - Rutgers; New Jersey Medical School; IOVS, Newark, New Jersey
  - Glaucoma Institute of Northern NJ, LLC, Rochelle Park, New Jersey
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Edward Harkness Eye Institute / Columbia University Medical Center, New York, New York
  - UNC Kittner Eye Center, Chapel Hill, North Carolina
  - Devers Eye Institute/Legacy Health, Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Robert Cizik Eye Clinic, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Eye Institute, Richmond, Virginia
  - University of Washington Medicine Eye Institute, Seattle, Washington
  - WVU Eye Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
To the American Glaucoma Society members after completion of the study, with an institutional review board (IRB) approved protocol.

REFERENCES:
- [Background] Arora KS, Robin AL, Corcoran KJ, Corcoran SL, Ramulu PY. Use of Various Glaucoma Surgeries and Procedures in Medicare Beneficiaries from 1994 to 2012. Ophthalmology. 2015 Aug;122(8):1615-24. doi: 10.1016/j.ophtha.2015.04.015. Epub 2015 Jun 16. PMID 26092196
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL; Tube versus Trabeculectomy Study Group. Treatment outcomes in the Tube Versus Trabeculectomy (TVT) study after five years of follow-up. Am J Ophthalmol. 2012 May;153(5):789-803.e2. doi: 10.1016/j.ajo.2011.10.026. Epub 2012 Jan 15. PMID 22245458
- [Background] Budenz DL, Barton K, Gedde SJ, Feuer WJ, Schiffman J, Costa VP, Godfrey DG, Buys YM; Ahmed Baerveldt Comparison Study Group. Five-year treatment outcomes in the Ahmed Baerveldt comparison study. Ophthalmology. 2015 Feb;122(2):308-16. doi: 10.1016/j.ophtha.2014.08.043. Epub 2014 Oct 17. PMID 25439606
- [Background] Anand A, Tello C, Sidoti PA, Ritch R, Liebmann JM. Sequential glaucoma implants in refractory glaucoma. Am J Ophthalmol. 2010 Jan;149(1):95-101. doi: 10.1016/j.ajo.2009.07.019. Epub 2009 Oct 17. PMID 19837382
- [Background] Burgoyne JK, WuDunn D, Lakhani V, Cantor LB. Outcomes of sequential tube shunts in complicated glaucoma. Ophthalmology. 2000 Feb;107(2):309-14. doi: 10.1016/s0161-6420(99)00039-1. PMID 10690831
- [Background] Ness PJ, Khaimi MA, Feldman RM, Tabet R, Sarkisian SR Jr, Skuta GL, Chuang AZ, Mankiewicz KA. Intermediate term safety and efficacy of transscleral cyclophotocoagulation after tube shunt failure. J Glaucoma. 2012 Feb;21(2):83-8. doi: 10.1097/IJG.0b013e31820bd1ce. PMID 21336148
- [Background] Jimenez-Roman J, Gil-Carrasco F, Costa VP, Schimiti RB, Lerner F, Santana PR, Vascocellos JP, Castillejos-Chevez A, Turati M, Fabre-Miranda K. Intraocular pressure control after the implantation of a second Ahmed glaucoma valve. Int Ophthalmol. 2016 Jun;36(3):347-53. doi: 10.1007/s10792-015-0125-z. Epub 2015 Sep 3. PMID 26334729
- [Background] Semchyshyn TM, Tsai JC, Joos KM. Supplemental transscleral diode laser cyclophotocoagulation after aqueous shunt placement in refractory glaucoma. Ophthalmology. 2002 Jun;109(6):1078-84. doi: 10.1016/s0161-6420(02)01019-9. PMID 12045047
- [Background] Smith M, Buys YM, Trope GE. Second Ahmed valve insertion in the same eye. J Glaucoma. 2009 Apr-May;18(4):336-40. doi: 10.1097/IJG.0b013e318182edfb. PMID 19365202
- [Background] Godfrey DG, Krishna R, Greenfield DS, Budenz DL, Gedde SJ, Scott IU. Implantation of second glaucoma drainage devices after failure of primary devices. Ophthalmic Surg Lasers. 2002 Jan-Feb;33(1):37-43. PMID 11820661
- [Background] Ko SJ, Hwang YH, Ahn SI, Kim HK. Surgical Outcomes of Additional Ahmed Glaucoma Valve Implantation in Refractory Glaucoma. J Glaucoma. 2016 Jun;25(6):e620-4. doi: 10.1097/IJG.0000000000000298. PMID 26091182
- [Background] Francis BA, Kawji AS, Vo NT, Dustin L, Chopra V. Endoscopic cyclophotocoagulation (ECP) in the management of uncontrolled glaucoma with prior aqueous tube shunt. J Glaucoma. 2011 Oct;20(8):523-7. doi: 10.1097/IJG.0b013e3181f46337. PMID 21048513
- [Background] Sood S, Beck AD. Cyclophotocoagulation versus sequential tube shunt as a secondary intervention following primary tube shunt failure in pediatric glaucoma. J AAPOS. 2009 Aug;13(4):379-83. doi: 10.1016/j.jaapos.2009.05.006. PMID 19683190
- [Background] Schaefer JL, Levine MA, Martorana G, Koenigsman H, Smith MF, Sherwood MB. Failed glaucoma drainage implant: long-term outcomes of a second glaucoma drainage device versus cyclophotocoagulation. Br J Ophthalmol. 2015 Dec;99(12):1718-24. doi: 10.1136/bjophthalmol-2015-306725. Epub 2015 May 29. PMID 26024673
- [Background] Gabelt BT, Kaufman PL. Changes in aqueous humor dynamics with age and glaucoma. Prog Retin Eye Res. 2005 Sep;24(5):612-37. doi: 10.1016/j.preteyeres.2004.10.003. PMID 15919228
- [Derived] Ma JX, Chuang AZ, Feldman RM, Mansberger SL, Tanna AP, Blieden LS, Shoham D, Bell NP, Gross RL, Pasquale LR, Greenfield DS, Liebmann JM, Weinreb RN; ASSISTS Study Group. Direct Costs of Second Aqueous Shunt Implant Versus Transscleral Cyclophotocoagulation (The Assists Trial). J Glaucoma. 2023 Mar 1;32(3):145-150. doi: 10.1097/IJG.0000000000002143. Epub 2023 Feb 1. PMID 36848258
- [Derived] Feldman RM, Chuang AZ, Mansberger SL, Tanna AP, Blieden LS, Bell NP, Gross RL, Pasquale LR, Greenfield DS, Liebmann JM, Weinreb RN; ASSISTS Group. Outcomes of the Second Aqueous Shunt Implant Versus Transscleral Cyclophotocoagulation Treatment Study: A Randomized Comparative Trial. J Glaucoma. 2022 Sep 1;31(9):701-709. doi: 10.1097/IJG.0000000000002079. Epub 2022 Jul 21. PMID 35901309

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 enrolled participants did not meet eligibility criteria and were excluded. Only one eye of each participant was eligible for enrollment.
Units Other Than Participants: eyes
Groups:
- Second Aqueous Shunt: Second Aqueous Shunt
  Either a Baerveldt Glaucoma Implant 350-mm2 BG101-350 or an Ahmed Model FP7 Flexible Plate must be used for all participants unless there is insufficient space, in which case a Baerveldt Glaucoma Implant 250-mm2 BG103-250 may be used.
  Baerveldt Glaucoma Implant 350-mm2 / BG101-350
  Ahmed Model FP7 Flexible Plate
  Baerveldt Glaucoma Implant 250-mm2 / BG103-250
Period: Overall Study
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Started | 23; 23 eyes | 22; 22 eyes
Randomized | 23; 23 eyes | 22; 22 eyes
Received Assigned Intervention | 22; 22 eyes | 20; 20 eyes
Week 1 Follow up | 22; 22 eyes | 19; 19 eyes
Month 1 Follow up | 22; 22 eyes | 18; 18 eyes
Month 3 Follow up | 21; 21 eyes | 18; 18 eyes
Month 6 Follow up | 19; 19 eyes | 19; 19 eyes
Month 12 Follow up | 16; 16 eyes | 16; 16 eyes
Year 2 Follow up | 6; 6 eyes | 9; 9 eyes
Year 3 Follow up | 7; 7 eyes | 5; 5 eyes
Completed | 7; 7 eyes | 5; 5 eyes
Not Completed | 16; 16 eyes | 17; 17 eyes
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 15 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (11.2) | 64.2 (9.8) | 63.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 16 | 13 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 8 | 17
  White | 11 | 9 | 20
  Other | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 20 | 42
Number of participants with hypertension [Count of Participants; unit: Participants] | 17 | 15 | 32
Number of participants with diabetes [Count of Participants; unit: Participants] | 9 | 8 | 17
Number of participants with autoimmune disease [Count of Participants; unit: Participants] | 3 | 1 | 4
Number of participants for whom study eye is right eye [Count of Participants; unit: Participants] | 15 | 5 | 20
Glaucoma type [Count of Participants; unit: Participants]
  Primary Open Angle | 9 | 10 | 19
  Primary Angle Closure | 1 | 1 | 2
  Mixed Open and Closed Glaucoma | 2 | 1 | 3
  Neovascular | 3 | 3 | 6
  Uveitis | 2 | 3 | 5
  Other Secondary Glaucoma | 5 | 2 | 7
Intraocular pressure (IOP) [Mean (Standard Deviation); unit: mmHg] | 27.6 (8.7) | 26.2 (9.7) | 26.9 (9.1)
Number of participants on ocular hypertensive medications [Count of Participants; unit: Participants] | 21 | 20 | 41
Number of ocular hypertensive medications per participant [Mean (Standard Deviation); unit: medications] | 3.2 (0.8) | 3.3 (1.1) | 3.2 (0.9)
Number of participants on oral carbonic anhydrase inhibitor (CAI) [Count of Participants; unit: Participants] | 2 | 4 | 6
Best corrected visual acuity as Assessed by the Snellen Chart Visual Acuity Test [Mean (Standard Deviation); unit: logMAR] — The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). Total score ranges from -0.3 logMAR to 1.4 logMAR, with a lower number indicating the ability to read smaller letters on the Snellen chart. A lower logMAR value indicates better visual acuity; a higher logMAR value indicates lower or poorer visual acuity.
  logMAR | 0.97 (0.90) | 0.49 (0.66) | 0.74 (0.82)

OUTCOME MEASURES:

1. Primary Outcome: Number of Eyes That Failed Treatment
Description: Treatment failure is defined as meeting one or more of the following 4 criteria:
  1. Intraocular pressure (IOP) a) >18 mm Hg on maximum tolerated topical IOP-lowering medications, or b) Reduction of < 20% IOP on maximum tolerated topical IOP-lowering medications from medicated preoperative IOP, or c) ≤ 5 mm Hg without IOP-lowering medications on IOP confirmation visit, 6 months after initial study intervention; or
  2. Reoperation for glaucoma; or
  3. Addition of an oral CAI for the study eye on or after the 6-Month Study Visit; or
  4. Loss of light perception vision (NLP).
Time Frame: from time of intervention to month 6
Population: Only one eye of each participant was eligible for enrollment. Data for this outcome measure were not collected for 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Number; unit: eyes
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
eyes | 0 | 0

2. Primary Outcome: Number of Eyes That Failed Treatment
Description: as for outcome 1
Time Frame: from month 6 to month 12
Population: Only one eye of each participant was eligible for enrollment. Data for this outcome measure were not collected for 4 in the Second Aqueous Shunt arm and 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Number; unit: eyes
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 18 | 19
eyes | 3 | 2

3. Primary Outcome: Number of Eyes That Failed Treatment
Description: as for outcome 1
Time Frame: from month 12 to year 3
Population: Only one eye of each participant was eligible for enrollment. Only those who did not fail treatment in the previous time period (previous time period is reported in Outcome measure 2) were analyzed in this time period. Data for this outcome measure were not collected for 15 in the Second Aqueous Shunt arm and 7 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Number; unit: eyes
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 7 | 13
eyes | 0 | 0

4. Secondary Outcome: Number of Eyes With Vision-threatening Complications
Time Frame: from the time of intervention to year 3
Population: as for outcome 1
Measure: Number; unit: eyes
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
eyes
  Hyphema | 2 | 0
  Hypotony persistent | 2 | 0
  Choroidal Effusion | 1 | 0
  Cystoid/Diabetic Macular Edema Progression | 2 | 3
  Primary Tube Complications | 2 | 0
  Cataract Progression | 0 | 3
  Macular Hole | 0 | 1
  Herpes Simplex Keratitis | 1 | 0
  Ectropion | 1 | 0
  Second Tube Migration Anteriorly | 1 | 0
  Vitreous Clogging Second glaucoma drainage device | 1 | 0
  Intraocular Lens Dislocation | 1 | 0
  Phacodonesis | 0 | 1

5. Secondary Outcome: Number of Eyes That Lost Two or More Lines of Vision as Assessed by the Snellen Chart Visual Acuity Test
Description: The Snellen visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). Loss of lines of vision indicates worsening visual acuity.
Time Frame: from time of intervention to year 3
Population: as for outcome 1
Measure: Number; unit: eyes
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
eyes | 3 | 8

6. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The week 1 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, week 1
Population: Data for this outcome measure was not collected 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
log MAgnification Requirement (logMAR) | 0.16 (0.45) | 0.14 (0.37)

7. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The month 1 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, month 1
Population: Data for this outcome measure was not collected for 5 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 15
log MAgnification Requirement (logMAR) | -0.03 (0.18) | 0.12 (0.20)

8. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The month 3 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, month 3
Population: Data for this outcome measure were not collected for 1 in the Second Aqueous Shunt arm and 3 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 21 | 17
log MAgnification Requirement (logMAR) | -0.10 (0.27) | 0.08 (0.13)

9. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The month 6 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, month 6
Population: Data for this outcome measure were not collected for 3 in the Second Aqueous Shunt arm and 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 19 | 19
log MAgnification Requirement (logMAR) | -0.03 (0.28) | 0.05 (0.30)

10. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The month 12 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, month 12
Population: Data for this outcome measure were not collected for 6 in the Second Aqueous Shunt arm and 4 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 16 | 16
log MAgnification Requirement (logMAR) | -0.06 (0.34) | 0.09 (0.31)

11. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The year 2 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, year 2
Population: Data for this outcome measure were not collected for 16 in the Second Aqueous Shunt arm and 11 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 6 | 9
log MAgnification Requirement (logMAR) | -0.28 (0.28) | 0.24 (0.46)

12. Secondary Outcome: Change in Visual Acuity as Assessed by the Snellen Chart Visual Acuity Test
Description: The visual acuity test is used to determine the smallest letters the participant can read on a standardized chart (Snellen chart). The year 3 reading minus the baseline reading is reported, with a positive number indicating a decrease in visual acuity (that is, an increase in logMAR value indicates a decrease in visual acuity).
Time Frame: baseline, year 3
Population: Data for this outcome measure were not collected for 16 in the Second Aqueous Shunt arm and 15 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: log MAgnification Requirement (logMAR)
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 6 | 5
log MAgnification Requirement (logMAR) | -0.23 (0.36) | 0.49 (0.76)

13. Secondary Outcome: Incidence of Pain
Description: Number of participants who reported pain.
Time Frame: 1 week
Population: Data for this outcome measure were not collected for 1 in the Second Aqueous Shunt arm and 2 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 21 | 18
Participants | 12 | 11

14. Secondary Outcome: Incidence of Pain
Description: Number of participants who reported pain.
Time Frame: 1 month
Population: Data for this outcome measure were not collected for 2 in the Second Aqueous Shunt arm and 2 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 20 | 18
Participants | 10 | 10

15. Secondary Outcome: Severity of Pain
Description: Severity of pain was assessed by the Universal Pain Assessment Tool, and the score ranges from 0 to 10, with a higher score indicating greater pain.
Time Frame: 1 week
Population: Data for this outcome measure were not collected for 1 in the Transscleral Cyclophotocoagulation arm and 2 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 21 | 18
score on a scale | 1.57 (1.99) | 1.44 (1.50)

16. Secondary Outcome: Severity of Pain
Description: as for outcome 15
Time Frame: 1 month
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 20 | 18
score on a scale | 1.40 (2.23) | 1.28 (1.36)

17. Secondary Outcome: Number of Office Visits Per Participant From Baseline to 3 Months
Time Frame: from baseline to 3 months
Population: Data for this outcome measure were not collected 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: office visits per participant
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
office visits per participant | 3.73 (2.53) | 0.95 (1.22)

18. Secondary Outcome: Number of Office Visits Per Participant Per Month After Month 3
Time Frame: from month 4 to year 3
Population: Data for this outcome measure were not collected for 2 in the Second Aqueous Shunt arm and 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: office visits per participant per month
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 20 | 19
office visits per participant per month | 0.35 (0.34) | 0.13 (0.14)

19. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute (NEI) Visual Function Questionnaire (VFQ) 25 (NEI-VFQ-25) - General Health Subscale
Description: The score on the National Eye Institute (NEI) Visual Function Questionnaire-25 (NEI-VFQ-25) subscale ranges from 0 to 100, with a higher score indicating greater functioning.
Time Frame: baseline
Population: Data for this outcome measure were not collected for 1 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 62.5 (21.5) | 48.7 (21.2)

20. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - General Health Subscale
Description: The score on the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) subscale ranges from 0 to 100, with a higher score indicating greater functioning.
Time Frame: month 12
Population: Data for this outcome measure were not collected for 8 in the Second Aqueous Shunt arm and 7 in the Transscleral Cyclophotocoagulation arm who received the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 58.9 (23.2) | 53.8 (20.0)

21. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - General Vision Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 64.5 (23.0) | 63.2 (15.3)

22. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - General Vision Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 64.3 (21.0) | 70.8 (22.5)

23. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Mental Health Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 55.4 (28.8) | 56.9 (30.0)

24. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Mental Health Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 57.6 (28.1) | 68.3 (30.0)

25. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Distance Activity Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 65.8 (24.2) | 63.5 (25.4)

26. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Distance Activity Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 75.8 (20.2) | 63.9 (28.1)

27. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Near Activity Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 66.3 (21.0) | 62.7 (20.5)

28. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Near Activity Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 71.2 (22.7) | 59.0 (27.3)

29. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Peripheral Vision Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 60.2 (24.0) | 59.2 (33.6)

30. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Peripheral Vision Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 62.5 (23.5) | 63.5 (33.3)

31. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Color Vision Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 86.4 (22.8) | 77.6 (26.2)

32. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Color Vision Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 91.1 (23.2) | 76.9 (25.9)

33. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Ocular Pain Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 76.2 (28.6) | 70.4 (16.3)

34. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Ocular Pain Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 83.0 (20.0) | 81.7 (19.5)

35. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Driving Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 63.1 (25.0) | 55.4 (13.7)

36. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Driving Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 56.5 (17.6) | 65.8 (14.9)

37. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Dependency Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 50.2 (22.5) | 46.7 (22.8)

38. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Dependency Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 49.3 (24.4) | 54.9 (23.2)

39. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Social Functioning Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 83.1 (18.7) | 82.7 (21.5)

40. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Social Functioning Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 83.3 (26.3) | 76.0 (34.8)

41. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Role Difficulty Subscale
Description: as for outcome 20
Time Frame: baseline
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 22 | 19
score on a scale | 54.8 (31.2) | 61.8 (26.8)

42. Secondary Outcome: Vision-related Quality of Life as Assessed by the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) - Role Difficulty Subscale
Description: as for outcome 20
Time Frame: month 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
Number analyzed (Participants) | 14 | 13
score on a scale | 63.4 (25.7) | 70.2 (31.7)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Second Aqueous Shunt | Transscleral Cyclophotocoagulation
All-Cause Mortality (participants affected / at risk) | 3/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 6/22 | 3/20
Other Adverse Events (participants affected / at risk) | 10/22 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Second Aqueous Shunt (N=22) | Transscleral Cyclophotocoagulation (N=20)
Death (General disorders) | 3 (3) | 0 (0)
Central Nervous System (CNS) Syphilis causing Pan Uveitis (Infections and infestations) | 1 (1) | 0 (0)
Left Lung Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyphema (Eye disorders) | 1 (1) | 0 (0)
Chest pain secondary to abdominal artery pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Acute on Chronic Combined Diastolic and Systolic Congestive Heart Failure exacerbation (Vascular disorders) | 1 (2) | 0 (0)
Left atrial myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pericardial effusion (Vascular disorders) | 1 (1) | 0 (0)
Purulent Constrictive Pericarditis, unspecified infectious etiology (Infections and infestations) | 1 (1) | 0 (0)
Heart Attack (Vascular disorders) | 0 (0) | 1 (1)
Non-ST-Elevation Myocardial Infarction (Vascular disorders) | 0 (0) | 1 (1)
Open Globe due to trauma (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Second Aqueous Shunt (N=22) | Transscleral Cyclophotocoagulation (N=20)
Acute on Chronic Respiratory Failure with Hypoxemia and Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Castochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Choroidals (Eye disorders) | 1 (1) | 0 (0)
Corneal Epithelial Defect (Eye disorders) | 1 (1) | 0 (0)
Decreased Visual Acuity (Eye disorders) | 2 (2) | 4 (4)
Development of Cystoid Macular Edema (Eye disorders) | 1 (1) | 1 (1)
Worsening of Cystoid Macular Edema (Eye disorders) | 0 (0) | 1 (1)
Dislipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic Macular Edema (Eye disorders) | 1 (1) | 1 (2)
Ectropion (Eye disorders) | 1 (1) | 0 (0)
Worsening Diabetic Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Filamentary Keratitis (Eye disorders) | 1 (1) | 0 (0)
Herpes Simplex Virus Dendritic Keratitis (Eye disorders) | 1 (1) | 0 (0)
Hyphema (Eye disorders) | 1 (1) | 0 (0)
Hypotony of eye (Eye disorders) | 1 (1) | 0 (0)
Leak/Inflammation or infection of eye (Infections and infestations) | 1 (1) | 0 (0)
Mild intraocular lens dislocation (inferior nasal) (Eye disorders) | 1 (1) | 0 (0)
Overfiltration of Eye (Eye disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (secondary) (Vascular disorders) | 1 (1) | 0 (0)
Re-exposed tube (Eye disorders) | 1 (1) | 0 (0)
Ssuperior nasal tube with <1 mm exposure at limbus (original tube) (Eye disorders) | 1 (1) | 0 (0)
Spot on gums (General disorders) | 1 (1) | 0 (0)
Throat Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Trabectome/Goniotomy of eye (Eye disorders) | 1 (1) | 0 (0)
Tube Migration Anteriorly (Eye disorders) | 1 (1) | 0 (0)
Vision loss from count fingers to light perception (Eye disorders) | 1 (1) | 0 (0)
Vitreous clogging of second tube shunt (Eye disorders) | 1 (1) | 0 (0)
Cataract formation (Eye disorders) | 0 (0) | 3 (3)
Worsening of cataract (Eye disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
No light perception (Eye disorders) | 0 (0) | 1 (1)
Phacodonesis (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT02691455/Prot_SAP_000.pdf